CLINICAL TRIAL: NCT03383276
Title: A Phase 1, Dose Escalating Study of the Safety, Tolerability, and Pharmacokinetics of IL-1-Ra Topically Administered to Eyes of Healthy Adult Subjects
Brief Title: Phase 1 Study for Safety and Tolerability of IL-1-Ra Topically Administered to Eyes of Healthy Adult Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Tongren Hospital (Other)
Collaborators: Chengdu Rhodiola Bio-Pharmaceutical Co Ltd (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2004L00946
Record Dates: First submitted 2017-12-19; First posted 2017-12-26 (Actual); Last update posted 2017-12-26 (Actual); Status verified 2017-12

CONDITIONS: Blepharokeratoconjunctivitis
MeSH Terms: interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IL-1Ra (Experimental)
  Interventions: Drug: IL-1Ra

INTERVENTIONS:
Drug: IL-1Ra — custom eye drop to be applied to the left eye.

SUMMARY:
The purpose of this study is to assess the safety and tolerability of ocular administration of Topical Interleukin-1-Receptor Antagonist in healthy volunteers. Additionally, the PK of Interleukin-1-Receptor Antagonist will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males and/or females between the ages of 18 and 45 years
* Medically healthy
* Best correction vision of greater than or equal to 20/20 in each eye
* BMI ≥ 19 and < 24 kg/m2
* Ability to understand and provide informed consent to participate in this study
* Willingness to follow study instructions and likely to complete all required visits

Exclusion Criteria:

* Any ocular or systemic diseases
* History of skin or ocular allergy symptoms
* Use contact lenses during the trails.
* Taking inhaled or oral steroids (for example Advair, Orapred)
* Have an active infection
* Have serologic evidence of HIV, Hepatitis C, Hepatitis C, or tuberculosis
* Receipt of any blood or blood products within 2 months prior to the first dosing day.
* Use any drugs within 2 weeks prior to the first dosing day.
* Use of cyclosporine, steroid eye drops, serum eye drops, or any other eye medication or experimental drug within the past 4 weeks.
* Have been exposed to an investigational drug/device within the preceding 3 months
* Pregnant or lactating females
* History of substance abuse, drug addiction or alcoholism
* Males and females unwilling to use an acceptable method of contraception for the duration of the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2017-12-18 (Actual); Primary Completion 2018-03-25 (Estimated); Study Completion 2018-06-10 (Estimated)

PRIMARY OUTCOMES:
Corneal fluorescein staining | 3 days
Best corrected visual acuity | 3 days
Ocular symptomatology | 3 days
Slit lamp examination | 3 days
Measurement of intraocularpressure | 3 days

SECONDARY OUTCOMES:
ELISA based assay to determine Pharmacokinetics for the evaluation of systemic exposure of IL-1Ra in healthy volunteers. | 3 days

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing TongRen Hospital, Beijing, China